CLINICAL TRIAL: NCT02089555
Title: Biomarkers for Alzheimer's Disease and Mild Cognitive Impairment in African Americans and Caucasians
Brief Title: African American Alzheimer's Progression Markers - CSF and Neuro-Imaging
Acronym: A3PM
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, William Hu MD/PhD, Assistant Professor of Neurology, Emory University
Other Study IDs: IRB00066145; R21AG043885 (NIH)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Spinal Puncture; Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, plasma, and DNA will be saved.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- African Americans: This group consists of African American (AA) individuals aged 65-80 who are part of the Emory Alzheimer's Disease Research Center (ADRC) (a multi-racial cohort of subjects with normal cognition, Mild Cognitive Impairment (MCI) or mild Alzheimer's Disease (AD)) or the Registry for Remembrance (RfR) (a community of AA individuals who are interested in studies of memory and aging). AA and Non-Hispanic White (NHW) participants will be frequency-matched for age, gender, and education within each cognitive category (35 with normal cognition, 30 with MCI, and 10 with mild AD for each race).
  Interventions: Procedure: Lumbar puncture; Procedure: Blood draw; Procedure: Magnetic Resonance Imaging (MRI)
- Non-Hispanic Whites: This group consists of Non-Hispanic White (NHW) individuals aged 65-80 who are part of the Emory Alzheimer's Disease Research Center (ADRC) (a multi-racial cohort of subjects with normal cognition, Mild Cognitive Impairment (MCI) or mild Alzheimer's Disease (AD)). African American (AA) and Non-Hispanic White (NHW) participants will be frequency-matched for age, gender, and education within each cognitive category (35 with normal cognition, 30 with MCI, and 10 with mild AD for each race).
  Interventions: Procedure: Lumbar puncture; Procedure: Blood draw; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Lumbar puncture — Cerebrospinal fluid (CSF) will be collected via lumbar puncture. During lumbar puncture, a needle is inserted between two lumbar bones (vertebrae) to remove a sample of cerebrospinal fluid. The procedure involves inserting a thin, hollow needle between the two lower vertebrae (lumbar region), through the spinal membrane (dura) and into the spinal canal and extracting a small amount of fluid. The procedure takes about 45 minutes.
  Other Names: Spinal tap
Procedure: Blood draw — One tube of blood will be collected in an ethylenediaminetetraacetic acid (EDTA)-K2 plasma tube for DNA analysis.
Procedure: Magnetic Resonance Imaging (MRI) — Each participant will undergo Magnetic Resonance Imaging (MRI) analysis using a modified Alzheimer's Disease Neuroimaging Initiative (ADNI) protocol with a 3 Tesla (3T) MRI Scan. The exam takes approximately 20 minutes.

SUMMARY:
African Americans are twice as likely to develop Alzheimer's disease as white Americans, but few African Americans are enrolled in large Alzheimer's biomarker studies. The current proposal aims to determine the influence of Alzheimer's disease and vascular disease on memory and aging in African Americans through modern biomarkers (spinal fluid, MRI, and amyloid imaging), and how these may differ between African Americans and white Americans in preparation for a large multi-center study of aging in African American.

DETAILED DESCRIPTION:
African Americans represent about 10% of the population in the US, but are under-represented in biomarker-related aging studies such as the Alzheimer's Disease Neuro-imaging Initiative (ADNI) and World Wide ADNI. Epidemiologic studies show that, compared to non-Hispanic white (NHW) Americans, African Americans (AA) are more likely to develop mild cognitive impairment (MCI) and Alzheimer's disease (AD), have different genetic risks of developing AD, and experience different rates of cognitive decline after cognitive symptoms develop. All these point to the existence of an MCI/AD endophenotype for AA, although few of these epidemiological studies involve modern chemical or imaging biomarkers associated with AD pathology and progression. Preliminary studies using AA subjects who have undergone CSF analysis (n=36) show that AA MCI subjects are more likely to have normal CSF AD biomarkers than NHW MCI subjects, yet at the same time greater hippocampal atrophy on MRI. The investigators hypothesize that endothelial dysfunction is an alternate mechanism which independently contributes to cognitive impairment in AA subjects with sub-threshold AD pathology in a race-independent fashion, and endothelia dysfunction further enhances the neurotoxicity of AD-associated brain changes in a race-dependent fashion. The investigators propose to build on their success in recruiting AA volunteers into memory and aging studies at the Emory's Registry for Remembrance to recruit a cross-sectional cohort of 75 AA subjects along with 75 NHW subjects with normal cognition, MCI, or mild AD. They will test this hypothesis through two aims. In Aim 1, they will determine whether endothelial dysfunctions independently contribute to cognitive decline in AA and NHW subjects by measuring cerebrospinal fluid (CSF) levels of AD, endothelial, and inflammatory markers. Each subject will also undergo MRI analysis for total area of white matter hyperintensities as an imaging marker of endothelial dysfunction. Based on the hypothesis, they predict that AA MCI/AD subjects are more likely than NHW MCI subjects to have normal CSF AD biomarkers, abnormal CSF endothelial markers, and greater number and area of white matter hyperintensities on MRI. In Aim 2, the investigators will determine if an endothelial marker - intercellular adhesion molecule 1 or ICAM-1 - gene variant unique to AA enhances AD neurotoxicity to explain the greater hippocampal atrophy among AA MCI subjects. The Lys56Met ICAM1 gene variant associated with low ICAM-1 levels is uniquely found in 16-20% of AA, and these subjects may have impaired downstream activation of neprilysin, an Abeta-degrading enzyme. If the hypothesis is true, AA subjects with the Lys56Met gene variant will be more likely to have hippocampal atrophy, temporal-parietal cerebral hypoperfusion, and cerebral amyloid deposition than AA subjects and NHW subjects without the gene variant. This may occur in the setting of CSF Abeta2 pseudo-normalization if low neprilysin levels lead to increased Abeta42 levels. Successful completion of the current proposal will confirm the preliminary finding of a unique AA endophenotype within the broader AD-spectrum disorders, directly examine whether endothelial dysfunctions additively and synergistically lead to cognitive decline in AD among AA in a cross-sectional cohort, and help power and design a future a multi-center, multi-racial longitudinal biomarker study to validate these cross-sectional findings.

ELIGIBILITY:
Inclusion Criteria:

* Ages 60-85.
* Has normal cognition, a diagnosis of mild cognitive impairment, or a diagnosis of Alzheimer's disease or mild cognitive impairment.
* Self-reported race of African American or non-Hispanic white.
* Able to undergo neuropsychological testing, lumbar puncture, and MRI.
* English speaking.

Exclusion Criteria:

* History of stroke.
* Diagnosis of Parkinson's disease, amyotrophic lateral sclerosis, or another progressive neurological disorder which may spare cognition.
* Mini-Mental State Examination (MMSE) < 17

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African American and non-Hispanic white seniors with normal cognition, mild cognitive impairment (MCI), or mild Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
CSF endothelial marker levels | one time only
CSF Alzheimer's biomarker levels | one time only

SECONDARY OUTCOMES:
MRI evidence of small vessel disease | one time only
MRI evidence of brain atrophy | one time only

CONTACTS AND LOCATIONS:
Overall Officials: William Hu, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Howell JC, Watts KD, Parker MW, Wu J, Kollhoff A, Wingo TS, Dorbin CD, Qiu D, Hu WT. Race modifies the relationship between cognition and Alzheimer's disease cerebrospinal fluid biomarkers. Alzheimers Res Ther. 2017 Nov 2;9(1):88. doi: 10.1186/s13195-017-0315-1. PMID 29096697
- See also: Emory Alzheimer's Disease Research Center — https://www.med.emory.edu/ADRC/